CLINICAL TRIAL: NCT02278744
Title: A Phase I Dose Escalation Trial for Salvage Re-Irradiation of Metastatic Spine Lesions Using Single-Fraction Stereotactic Radiosurgery
Brief Title: Trial for Salvage Re-Irradiation of Metastatic Spine Lesions Using Single-Fraction Stereotactic Radiosurgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-054
Record Dates: First submitted 2014-10-27; First posted 2014-10-30 (Estimated); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Spine Lesions
Keywords: Single-Fraction Stereotactic Radiosurgery; Salvage Re-Irradiation; 14-054
MeSH Terms: interventions — Radiosurgery

ARMS (1):
- single-fraction radiosurgery (Experimental)
  Interventions: Radiation: single-fraction radiation; Device: MRI and/or CT

INTERVENTIONS:
Radiation: single-fraction radiation — Patients enrolled on this study will be registered into a dose tier and undergo 1 session of image-guided SRS using techniques previously. Three escalating SRS spinal cord/cauda maximum dose (Dmax) levels (14 Gy, 16 Gy, and 17 Gy) will be evaluated to determine the safety of this approach. A minimum of three patients will be treated per dose tier. Toxicity based on NCI CTCAE (v4). Post treatment followup at 2 and 4 months (+/- 2 weeks) post-treatment, at 6 months (+/- 4 weeks) and then every 3 months until 2 years (± 4 weeks). Followup schedule based on last day of treatment. No schedule adjustments based on early or delayed visits.
  Other Names: stereotactic radiosurgery (SRS)
Device: MRI and/or CT

SUMMARY:
This is a phase I clinical trial investigating the use of single fraction re-irradiation following local progression of spine and cauda equina (L2 to sacrum) lesions that have previously received radiation therapy. Patients will be treated with single-fraction radiation therapy at 3 dose levels using image-guided stereotactic radiosurgery techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic or cytologic proof of a non-hematologic malignancy confirmed by MSKCC pathologic review
* Patients must have radiographic evidence of malignancy in the spine or cauda equina region (L2 to sacrum) which is suitable for radiation therapy
* Patients must have received prior external beam radiation therapy to the region proposed for SRS re-irradiation at least 6 months prior to planned re-irradiation
* For patients who were previously treated at an outside institution, adequate records must be available to determine the true dose the cord/cauda received during prior RT. Sufficiency of the treatment records will be assessed and signed-off by the Medical Physics investigator.
* Patients must have demonstrated progression of disease on MRI or CT assessment of the spinal cord/cauda within the previous radiation field

  o progression may consist of an increase in maximal dimension of the tumor by ≥20%, compromise of the spinal cord/cauda equina and/or exiting spinal nerves (assessed clinically or radiographically), or both.
* Target lesion size for re-irradiation must be ≤ 2 vertebral bodies
* KPS ≥ 60%
* Age ≥ 18 years old

Exclusion Criteria:

* Patients with a life expectancy of < 6 months as predicted by the Adult Comorbidity Index (ACE-27, see Appendix 1).
* Patients with intradural or intramedullary lesions, or lesions with < 2mm distance from tumor to spinal cord
* Patients with circumferential epidural disease
* Systemic chemotherapy delivered or planned to be delivered within (+/-) 5 days of SRS re-irradiation
* Patients receiving bevacizumab within 12 weeks prior to protocol treatment.
* Unable to undergo either a myelogram or MRI of spinal cord/cauda equina and/or exiting spinal nerves
* Patients who may not receive therapeutically effective doses via an external beam approach to the lesion of interest as specified by the Dose Limit Guidelines Evaluation of doses previously delivered to spinal cord/cauda equina and other critical structures (bowel, esophagus, kidneys, rectum) will be taken into consideration

  * If repeat irradiation would exceed any normal tissue constraint as noted in Appendix 2, the patient will be ineligible
  * If the total prior radiation dose to the spinal cord/cauda equina and/or sacrum over all prior treatments exceeds 100 Gy BED (biologically effective dose), the patient will be ineligible, where a total of 100 Gy BED is determined by the calculation: BED = nd(1 + d/α/β), where n = number of fractions and d = dose per fraction; α/β is the constant for spinal cord/cauda/sacrum late effect and equals 2 [Rades 2005, Nieder 2005, Sahgal 2012]
* Patients with paraspinal extension of disease with visceral involvement exclusive of patients with cauda equina and sacral disease extension.
* Abnormal complete blood count. Any of the following:

  * Platelet count < 75,K/mcL
  * Hemoglobin level < 9g/dl
  * WBC < 3.5K/mcL
* Abnormal coagulation profile: INR > 2.5 and/or PTT > 80

  o Patients who are on anticoagulation medication that may not be safely held for the procedure (≥ 5 days for antiplatelet agents and warfarin; ≥ 24 hours for low-molecular weight heparin formulations) will be excluded
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
toxicities as measured by the National Cancer Institute (NCI) Common Toxicity Criteria | 1 year
  The toxicities associated with single fraction stereotactic radiosurgery to the spine may be classified as either early (occurring within 90 days of the treatment) or late toxicities (after 90 days to 1 year). These toxicities will be evaluated with the National Cancer Institute (NCI) Common Toxicity Criteria.

SECONDARY OUTCOMES:
local failure | 1 year
  tumor control will be defined for this study as the absence of tumor progression at the treated site, where progression may consist of an increase in maximal dimension of the tumor by ≥20%, compromise of the spinal cord/cauda equina and/or exiting spinal nerves (assessed clinically or radiographically), or both.
overall survival | 2 years
  will be evaluated from the completion of treatment, and analyzed by the Kaplan-Meier method or cumulative incidence curves. For these outcomes, patients across all dose levels will be combined, and will only be evaluated for a maximum of 2 years on protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiya Yamada, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/